CLINICAL TRIAL: NCT01607346
Title: An Open Label Study to Evaluate the Effects of Ezogabine/Retigabine Added to Existing Anti-epileptic Drug(s) on Urinary Voiding Function in Subjects With Partial Onset Seizures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116158; 2012-002260-26 (EudraCT Number)
Record Dates: First submitted 2012-05-17; First posted 2012-05-30 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Epilepsy
Keywords: Urinary Retention
MeSH Terms: conditions — Epilepsy; Urinary Retention | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ezogabine/retigabine (Experimental): Open-label
  Interventions: Drug: ezogabine/retigabine

INTERVENTIONS:
Drug: ezogabine/retigabine — Starting dose of 300mg/day, titrate up to a targeted maximum dose of 1200 mg/day. Dose can be reduced to a minimum of 600 mg/day if unable to tolerate higher doses

SUMMARY:
This is a multicentre, open label study to examine the effect of ezogabine/retigabine on the voiding function of adult subjects with drug-resistant partial onset seizures (POS). Subjects fulfilling the study entry criteria at Screening and at Baseline including a comprehensive eye examination by an ophthalmologist or retina specialist and a skin assessment by the investigator will receive ezogabine/retigabine.

The starting dose of ezogabine/retigabine will be 300 mg/day. Subjects will be up titrated by 150 mg/day weekly up to the maximum ezogabine/retigabine daily dose of 1200 mg (or the highest tolerated dose). During the 49 days of the treatment phase, subjects will undergo three repeat non-invasive assessments of voiding function. In addition, subjects who meet pre-determined criteria for voiding dysfunction will undergo multichannel cystometry in order to characterise bladder hypocontractility, bladder outlet obstruction or a combination of events which clinically is manifest with difficulty emptying the bladder or acute urinary retention.

At the end of the Treatment Phase, all subjects will enter the Taper Phase, a 3-week down titration period. Subjects who have new findings of abnormal pigmentation of the retina, unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of skin, lip, nail, or mucosa since baseline will be asked to enter the Safety Follow-Up / Continuation Phase. All subjects will undergo 6-monthly comprehensive eye examinations during the Safety Follow-Up / Continuation Phase. Subjects who have not developed abnormal discoloration of the skin, lips, nails or mucosa will continue to undergo skin assessments by the investigator. Any subject who has developed abnormal discoloration of the skin, lips, nails or mucosa since baseline will be referred to a dermatologist for evaluation and 6-monthly follow up assessments. All subjects will continue to be followed until the pigmentation and/or discoloration has resolved or stabilised, as defined by no change over 2 consecutive 6-monthly assessments conducted over at least 12 months after discontinuation of ezogabine/retigabine.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥18 years of age (male or female).
* Has a confident diagnosis of epilepsy with partial onset seizures with or without secondary generalization (classified according to International League Against Epilepsy (ILAE) Guidelines, 1981) ≥ 2 years.
* Is currently being treated with a stable regimen of one to three AEDs during the 4 weeks prior to the Screening Visit.
* Following Amendment 03: must be considered drug resistant, consistent with the definition proposed by Kwan, et al 2010 [Kwan].
* Note: Vagus Nerve Stimulator (VNS), VNS will not be counted as a concurrent AED. Subjects with surgically implanted VNS will be allowed to enter the study provided that all of the following conditions are met:
* The VNS has been in place for at least 24 weeks prior to the Screening Visit
* The settings must remain the same for at least 4 weeks prior to the Screening Visit and throughout the study
* The battery is expected to last for the duration of the study
* Subject who are considering implantation of a VNS are excluded from participating in this study
* Note: The chronic use of benzodiazepines as a concurrent AED is permitted as long as the dose is kept constant for at least 4 weeks before the Screen Visit and throughout the study.
* Is able and willing to maintain an accurate and complete a two (2) day Voiding Diary at protocol specified time points.
* Is able and willing to maintain an accurate and complete daily written Seizure Calendar at specified time points or has a caregiver who is able and willing to maintain an accurate and complete daily written Seizure Calendar for the entire duration of the study.
* Has given written informed consent, prior to the performance of any study assessments.
* A female subject is eligible to enter and participate in the study if she is not pregnant or lactating or planning to become pregnant during the study and is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal).
* Pre-menopausal females with a documented (medical report verification) hysterectomy with or without oophorectomy or bi-lateral oophorectomy when reproductive status has been confirmed by hormone level assessment
* Post-menopausal females defined as being amenorrhoeic for greater than one year with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms). However, if indicated, this should be confirmed by oestradiol and follicle stimulating hormone (FSH) levels consistent with menopause (according to local laboratory ranges).
* Women who have not been confirmed as post-menopausal should be advised to use contraception as outlined in Appendix 2.
* Child-bearing potential, has a negative pregnancy test at screening and baseline, and agrees to satisfy one of the requirements in as listed in Appendix 2.
* Liver function tests: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2 x upper limit of normal (ULN); alkaline phosphatase and bilirubin less than or equal to 1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Has a normal creatinine clearance (age corrected) as calculated with the Cockcroft-Gault formula.

Exclusion Criteria:

* Has generalized epilepsy (e.g., Lennox-Gastaut, Juvenile Myoclonic epilepsy, Absence, etc).
* Has had status epilepticus (other than simple partial status epilepticus) within the 12 months prior to Screening or during the Baseline Phase.
* Has a history of innumerable seizures within the 12 months prior to Screening where the individual seizures cannot be counted.
* Has a history of pseudo seizures, non-epilepsy events or any other type of psychogenic seizures that could be confused with seizures.
* Acute Urinary Retention (treated or untreated) within 6 months of screening or an episode of Acute Urinary Retention (treated) within the last two years with symptoms within the last 6 months.
* Screening AUA SI Score >7 (>11 for subject over 55 years old).
* Flowmetry Peak Flow < 15mL/sec out of a urine volume void of 150mL (<11 mL/sec for subject over 55 years old) at Screening.
* PVR >125mL or >40% functional residual volume at Screening.
* Prior history of administration of Botox® within genitourinary system.
* Prior history or any type of medical or surgical therapy for urinary incontinence.
* Prior history of treated or untreated, bladder, prostate, uterine or cervical cancer.
* Use of sildenafil, tadalafil, vardenafil or other PDE-5 inhibitors within 2 weeks of study start.
* Use of α-adrenoreceptor antagonists within 2 weeks of study start.
* Has had previous exposure to ezogabine/retigabine.
* Is currently or has been abusing substance(s) or any medications in the 12 months prior to Screening.
* Has taken an investigational drug, or used an investigational device, within the previous 4 weeks prior to Screening or plans to take another investigational drug anytime during the study.
* Is currently following or planning to follow the ketogenic diet.
* Has been treated with felbamate or vigabatrin within the past 6 months prior to Screening; if a subject has been previously treated with vigabatrin, a visual perimetry test prior to screening (or within the past 6 months) must show normal visual fields or no worsening of recognized visual field abnormalities as compared with prior to vigabatrin treatment.
* Use of CNS-active medication (other than concomitant AED therapy), unless subjects had been stabilized on such medication for more than 4 weeks prior to Screening.
* Use of herbal treatments with CNS activity within 4 weeks prior to Screening.
* Current use of any prohibited concomitant medication as indicated in Section 5.7.2.
* Is planning surgery to control seizures during the study.
* Is suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormalities that, in the investigator's judgment, are likely to interfere with the objectives of the study.
* Has any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome, including but not limited to: clinically significant cardiac, renal, hepatic condition, or a condition that affects the absorption, distribution, metabolism or excretion of drugs.
* Has an average QTc ≥ 450 msec or ≥ 480 msec for subjects with Bundle Branch Block at the time of Screening.

Note: If the initial electrocardiogram (ECG) at Screening indicates a corrected QT (QTc) interval outside these limits, two further ECGs should be performed and the average QTc value of these triplicate ECGs calculated. If the average value exceeds the stated limits, the subject is not eligible.

* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than one lifetime suicide attempt.
* Has positive test results for hepatitis B surface antigen, positive hepatitis C virus, or human immunodeficiency virus (HIV)-1 or -2 at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Madison, Wisconsin
- France (2):
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Strasbourg
- GSK Investigational Site, Warsaw, Poland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, open label study to examine the effect of ezogabine/retigabine added to existing anti-epileptic drugs on the voiding function of adult participants with drug-resistant partial onset seizures (POS). The study was conducted in two countries: United States and France.
Pre-assignment Details: The study was conducted in 5 phases:Screening (Day-30 to Day-2), Baseline (Day-1), treatment (Day1-49), taper-down titration (Day 50-70). A total of 10 participants were enrolled into the study and received at least one dose of the study medication.
Groups:
- Ezogabine/Retigabine: Participants received ezogabine/retigabine tablets orally in three equally divided doses each day with or without food. The starting dose of ezogabine/retigabine was 300 milligrams (mg)/day. Participants were to be up titrated by 150 mg/day weekly up to a minimum ezogabine/retigabine daily dose of 600 mg/day and a maximum ezogabine/retigabine daily dose of 1200 mg/day. If participants missed one dose or more, it was recommended that they took a single dose as soon as they remember. After taking a missed dose, at least 3 hours were to elapse before the next dose and then the normal dosing schedule was to be resumed. After Day 22 of treatment, if a participant was unable to tolerate doses of ezogabine/retigabine greater than 600 mg/day, the investigator was able to decrease the dose as appropriate.
Period: Overall Study
Arm/Group | Ezogabine/Retigabine
Started | 10
Completed | 7
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum Flow Rate (Qmax) at Visit 5.
Description: Maximum urine flow rate was measured by uroflowmetry test. It is a non-invasive diagnostic test that measures the speed of urinary flow. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visits 3, 4 and 5 (Days 21, 35 and 49 respectively). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value at Visit 5. Safety Population was defined as all participants who received more than or equal to one dose of study medication.
Time Frame: Baseline (Day -1) and on Day 49 (Visit 5)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter (mL) per second
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 7
Milliliter (mL) per second | -1.49 (4.797)

2. Secondary Outcome: Change From Baseline in Maximum Flow Rate (Qmax) at Visits 3, 4 and 6
Description: Maximum urine flow rate was measured by uroflowmetry test. It is a non-invasive diagnostic test that measures the speed of urinary flow. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visits 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL per second
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
mL per second
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | -5.32 (5.669)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | -3.83 (9.796)
  Visit 6, n=10 | -2.22 (6.742)

3. Secondary Outcome: Percent Change From Baseline in Qmax at Visits 3, 4, 5 and 6
Description: Maximum urine flow rate was measured by uroflowmetry test. It is a non-invasive diagnostic test that measures the speed of urinary flow. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visits 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. The percentage change from Baseline was calculated as post-baseline value minus Baseline value divided by Baseline value multiplied by 100. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Percent change
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | -23.45 (22.444)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | -6.53 (38.253)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | -1.44 (18.800)
  Visit 6, n=10 | -7.14 (27.743)

4. Secondary Outcome: Change From Baseline in Percentage Residual Urinary Volume (RUV) at Visits 3, 4, 5 and 6
Description: Percentage residual urinary volume is a standardized measure of post-residual volume and is defined as residual devided by residual plus voided multiplied by 100 where 'residual' is the post-void residual (PVR) volume collected on the bladder ultrasound and 'voided' is the voided volume collected on the uroflowmetry. Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated as post-baseline minus Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of residual urinary volume
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Percentage of residual urinary volume
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | 1.09 (17.450)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | 3.77 (15.167)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | -0.18 (19.716)
  Visit 6, n=10 | 7.56 (18.253)

5. Secondary Outcome: Change From Baseline in Voided Volume (VV) at Visits 3, 4, 5 and 6
Description: The volume of urine voided was measured by uroflowmetry test. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visits 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
mL
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | -81.3 (208.21)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | -96.8 (205.80)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | 37.6 (225.33)
  Visit 6, n=10 | -68.9 (164.20)

6. Secondary Outcome: Change From Baseline in Time to Maximum Flow at Visits 3, 4, 5 and 6
Description: Time to maximum flow was measured by uroflowmetry test. It is a non-invasive diagnostic test that measures the speed of urinary flow. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visits 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Seconds
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | 2.80 (6.588)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | 3.63 (12.683)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | 6.51 (11.476)
  Visit 6, n=10 | -1.78 (6.296)

7. Secondary Outcome: Change From Baseline in Flow Time at Visits 3, 4, 5 and 6
Description: Flow time was measured by uroflowmetry test. It is a non-invasive diagnostic test that measures the speed of urinary flow. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visit 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Seconds
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | 0.22 (10.269)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | -1.13 (6.873)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | 9.07 (14.007)
  Visit 6, n=10 | -1.63 (12.278)

8. Secondary Outcome: Change From Baseline in Average Flow Rate (Qmean) at Visits 3, 4, 5 and 6
Description: Average flow rate was measured by uroflowmetry test. It is a non-invasive diagnostic test that measures the speed of urinary flow. Uroflowmetry was assessed at Baseline visit 2 (Day -1) and on visit 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL per second
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
mL per second
  Visit 3, n=9: number analyzed (Participants) | 9
  Visit 3, n=9 | -1.97 (5.406)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | -2.80 (7.085)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | -1.04 (4.295)
  Visit 6, n=10 | -2.62 (5.765)

9. Secondary Outcome: Frequency of Micturition as Recorded on the Voiding Diary for 2 Days Prior to Each Visit
Description: The participants were asked to complete a voiding diary for two days preceding each visit. Frequency of micturition for 2 days prior to dach visit was defined as total number of entries recorded within 2 days prior to each post-baseline visit. Voiding diary was assessed at Baseline visit 2 (Day -1) and on visit 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micturition voided
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Micturition voided
  Visit 3, n=8: number analyzed (Participants) | 8
  Visit 3, n=8 | 8.1 (3.60)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | 9.4 (5.32)
  Visit 5, n=6: number analyzed (Participants) | 6
  Visit 5, n=6 | 9.7 (4.72)
  Visit 6, n=9: number analyzed (Participants) | 9
  Visit 6, n=9 | 9.7 (5.27)

10. Secondary Outcome: Volume Voided as Recorded on the Voiding Diary for 2 Days Prior to Each Post-baseline Visit
Description: The participants were asked to complete a voiding diary for two days preceding each visit. Volume voided for 2 days prior to each visit was defined as sum of urine recorded within 2 days prior to each post-baseline visit. Voiding diary was assessed at Baseline visit 2 (Day -1) and on visit 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
mL
  Visit 3, n=8: number analyzed (Participants) | 8
  Visit 3, n=8 | 2850.1 (1238.42)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | 3558.1 (1713.81)
  Visit 5, n=6: number analyzed (Participants) | 6
  Visit 5, n=6 | 3470.8 (1463.08)
  Visit 6, n=9: number analyzed (Participants) | 9
  Visit 6, n=9 | 2736.1 (1466.70)

11. Secondary Outcome: Change From Baseline in American Urological Association Symptom Index (AUA SI) at Visits 3, 4, 5 and 6
Description: The America Urological Association Symptom Index is a 7-item Likert-scored scale describing urinary bladder function. It is the sum of the responses to the 7 AUA symptom questions. Score ranges from 0 to 5 (0=not at all and 5=almost always for questions 1 to 6; 0=None and 5=five times or more for question 7). The total score ranges from 0-35 where higher scores indicate more severe symptoms. It was completed by the investigator at Baseline visit 2 (Day -1) and on visit 3 (Day 21), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Measurement at visit 2 (Day -1) was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Day -1) and up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
Scores on a scale
  Visit 3, n=10 | 1.6 (3.10)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | 0.7 (1.25)
  Visit 6, n=10 | 0.4 (1.51)

12. Secondary Outcome: Cystometry Assessment at Visits 3, 4, 5 and 6
Description: Cystometry is a test of bladder function in which pressure and volume of fluid in the bladder is measured during filling, storage, and voiding. Cystometry was assessed at Baseline visit 2 (Day -1) and on visit 3 (Day 21), visit 4 (Day 35), visit 5 (Day 49) and visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). The requirement for cystometry was discovered by the study monitor and discussed with the GSK medical monitor after the participants had completed the study.
Time Frame: Up to Day 80 (Visit 6)
Population: Data were not collected, although 3 participants met at least 1 of the criteria for multichannel cystometry during the study, the assessment was not performed.
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in PVR Volume by Bladder Ultrasound at Visits 3, 4, 5 and 6
Description: PVR is the the amount of urine left in the bladder after urination. Bladder ultrasound was performed to assess PVR at Baseline/Visit 2 (Day -1), Visit 3 (Day 21), Visit 4 (Day 35), Visit 5 (Day 49) and Visit 6 (follow-up visit within 14 days after the end-of-treatment eye examination). Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 80 (Visit 6)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 10
mL
  Visit 3, n=10 | -17.2 (88.05)
  Visit 4, n=8: number analyzed (Participants) | 8
  Visit 4, n=8 | -6.3 (88.00)
  Visit 5, n=7: number analyzed (Participants) | 7
  Visit 5, n=7 | -13.9 (105.67)
  Visit 6, n=10 | 3.5 (64.09)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of the study treatment until the follow-up visit within 14 days after the end-of-treatment eye examination (approximately up to 80 days).
Description: On treatment SAEs and non-serious AEs were reported for the Safety Population which included all participants who received more than or equal to one dose of study medication.
Arm/Group | Ezogabine/Retigabine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezogabine/Retigabine (N=10)
Ataxia (Nervous system disorders) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezogabine/Retigabine (N=10)
Palpitations (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Discomfort (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Oedema (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (6)
Dysarthria (Nervous system disorders) | 1 (2)
Paraesthesia (Nervous system disorders) | 2 (3)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Libido decreased (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated after 10 of 100 subjects had been enrolled. Statistical analyses were not performed as the sample size enrolled was too small to allow for these analyses to be meaningful. The data are presented as summary statistics only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.